CLINICAL TRIAL: NCT01823913
Title: Safety and Pharmacokinetic Comparison of Exforge® and G-0081 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Kyungsoo Park, Associate Professor, Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G-0081
Record Dates: First submitted 2013-03-24; First posted 2013-04-04 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
Keywords: Pharmacokinetics

ARMS (1):
- Test and reference formulations (Experimental): Test formulation and reference formulation given orally 14 days apart in a fasted state
  Interventions: Drug: Test formulation; Drug: Reference formulation

INTERVENTIONS:
Drug: Test formulation — A single oral dose of a combination tablet of amlodipine orotate 10mg and valsartan 160mg
Drug: Reference formulation — A single oral dose of a combination tablet of amlodipine besylate 10mg and valsartan 160mg

SUMMARY:
This study investigates safety and pharmacokinetic comparison of G-0081, a combination tablet of amlodipine and valsartan (test formulation), and Exforge®, a combination tablet of amlodipine and valsartan (reference formulation) for single dose in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers between the ages of 20 and 50 and within 20% of their ideal body weight, without congenital abnormality or chronic disease

Exclusion Criteria:

* History of cardiovascular, pulmonary, renal, endogenous, gastrointestinal, hematologic, neurologic or hemorrhagic disease;
* Clinically significant findings on routine laboratory (hematology, serum chemistry and urinalysis) or ECG tests;
* Use of prescription drugs in the 14 days immediately prior to starting the study that had the potential to interact with the study medication;
* Use of any substance that could induce or inhibit drug metabolism enzymes

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Profile of Pharmacokinetics | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 144, 192 hours post-dose
  Cmax, Area Under Curve(0 to the last sampling time)

SECONDARY OUTCOMES:
Profile of Pharmacokinetics | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 144, 192 hours post-dose
  Tmax, Area Under Curve(0 to infinity), T_1/2

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim Y, Son M, Lee D, Roh H, Son H, Chae D, Bahng MY, Park K. Pharmacokinetic comparison of 2 fixed-dose combination tablets of amlodipine and valsartan in healthy male Korean volunteers: a randomized, open-label, 2-period, single-dose, crossover study. Clin Ther. 2013 Jul;35(7):934-40. doi: 10.1016/j.clinthera.2013.05.021. PMID 23870605